CLINICAL TRIAL: NCT05984212
Title: Effect of Preoperative Rectus Sheath Block on Quality of Recovery in Single Port Laparoscopic Adnexal Surgery: A Randomized Controlled Trial
Brief Title: Effect of Preoperative Rectus Sheath Block on Quality of Recovery in Single Port Laparoscopic Adnexal Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 4-2023-0611
Record Dates: First submitted 2023-07-16; First posted 2023-08-09 (Actual); Last update posted 2023-08-09 (Actual); Status verified 2023-08

CONDITIONS: Single Port Laparoscopic Adnexal Surgery
MeSH Terms: interventions — Dexmedetomidine; Saline Solution

STUDY DESIGN:
Intervention Model Description: Double blind randomized controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Investigator prepared the drug and participant and outcomes assessor were blind to the group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dexmedetomidine infusion group (Experimental)
  Interventions: Drug: Ultrasound guided rectus sheath block with dexmedetomidine
- normal saline infusion group (Placebo Comparator)
  Interventions: Drug: Ultrasound guided rectus sheath block with normal saline

INTERVENTIONS:
Drug: Ultrasound guided rectus sheath block with dexmedetomidine — Intervention Group: Ultrasound guided rectus sheath block with 0.5% ropivacaine 20ml at each side (bilateral)
  Arms: dexmedetomidine infusion group
Drug: Ultrasound guided rectus sheath block with normal saline — Control Group: Ultrasound guided rectus sheath block with 0.9% normal saline 20ml at each side (bilateral)
  Arms: normal saline infusion group

SUMMARY:
In this study, the investigators aimed to demonstrate if the quality of recovery in patients undergoing single-port laparoscopic adnexal surgery, with preoperative rectus sheath block and intraoperative opioid administration based on analgesia nociception index, improves compared to the patients without block.

ELIGIBILITY:
Inclusion Criteria:

1. Adult female patient aged 19 years or older undergoing elective single-port laparoscopic adnexal surgery under general anesthesia at Yonsei Cancer Center

1. patients with moderate to severe pain before surgery 2. patients with history of taking chronic analgesic use, 3. patients allergic or hypersensite to remifentanil or local anesthetic (ropivacaine), 4. patients with infection at the site of the block, 5. patietns who cannot communicate

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Estimated)
Dates: Start 2023-08 (Estimated); Primary Completion 2024-07 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Quality of Recovery 40 scale score at postoperative 24 hour | 24 hours after the end of surgery
  Postoperative quality of recovery according to the block performance

SECONDARY OUTCOMES:
Intraoperative remifentanil consumption,postoperative pain score | at 0, 1, 6, 12, and 24 hours postoperative
  To evaluate the effect of rectus sheath block on intraoperative and postoperative pain and patients' satisfaction
rescue analgesics administered up to 24 hours postoperatively | intraoprative and postoperative 24hours
  To evaluate the effect of rectus sheath block on intraoperative and postoperative pain and patients' satisfaction
satisfaction with pain control | intraoprative and postoperative 24hours
  Patient self-rated overall satisfaction with pain control. Evaluated on an 11-point scale from 0 to 10, with 0 points for completely dissatisfied and 10 points for complete satisfaction. The higher the number, the more satisfactory it is.
serum cortisol level (μg/dL) before and after surgery | intraoprative and postoperative 24hours
  To evaluate the effect of rectus sheath block on intraoperative and postoperative pain and patients' satisfaction
leukocyte level (10^3/μL) before and after surgery | intraoprative and postoperative 24hours
  To evaluate the effect of rectus sheath block on intraoperative and postoperative pain and patients' satisfaction
arterial pH before and after surgery | intraoprative and postoperative 24hours
  To evaluate the effect of rectus sheath block on intraoperative and postoperative pain and patients' satisfaction
blood glucose level (mg/dL) before and after surgery | intraoprative and postoperative 24hours
  To evaluate the effect of rectus sheath block on intraoperative and postoperative pain and patients' satisfaction
measurement of adequate analgesia (NRS <4) before and after surgery | intraoprative and postoperative 24hours
  To evaluate the effect of rectus sheath block on intraoperative and postoperative pain and patients' satisfaction

CONTACTS AND LOCATIONS:
Overall Officials: Youngwon Kim, Principal Investigator — Department of Anesthesiology and Pain Medicine, Anesthesia and Pain Research Institute, Yonsei University College of Medicine
Locations (1):
- Severance hospital, Seoul, South Korea